CLINICAL TRIAL: NCT02207075
Title: Measuring Active Microglia in Progressive Multiple Sclerosis
Status: Completed | Type: Observational
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Other Study IDs: 1309014365
Record Dates: First submitted 2014-07-30; First posted 2014-08-01 (Estimated); Last update posted 2022-01-18 (Actual); Status verified 2022-01

CONDITIONS: Secondary Progressive Multiple Sclerosis
Keywords: SPMS; Myelin Water Fraction; activated microglia
MeSH Terms: conditions — Multiple Sclerosis, Chronic Progressive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Subjects with SPMS: Secondary progressive MS Subjects either untreated or on consistent treatment for six months prior to enrollment.
  SPMS subjects will have two baseline [11C]PK-11195 PET scans (separated by 24 to 72 hours, test-retest) and subsequent scans at 6, 12 and 24 months. SPMS Subjects will have brain MRI's at baseline, 6, 12 and 24 months.
  Interventions: Drug: [C11]PK-1195 PET scan
- Normal Control Subjects: Healthy Controls will have 2 baseline [C11]PK-1195 PET scans and 1 MRI.
  Interventions: Drug: [C11]PK-1195 PET scan

INTERVENTIONS:
Drug: [C11]PK-1195 PET scan — PET scan with tracer [C11]PK-1195

SUMMARY:
This is pilot study designed to quantifying the innate immune inflammatory burden in a cohort of secondary progressive multiple sclerosis subjects. Innate immunity is recognized as a major cause of tissue injury in central nervous system (CNS) disease. Our hypothesis is that the innate immune response is heightened in SPMS as compared to healthy controls (HC's) and this activity increases over time and correlates with ongoing neuronal loss and disability. The investigators will test this hypothesis by using highly specific molecular imaging techniques, specifically PET, in conjunction with high field MRI. The investigators will utilize the PET radioligand [11C]PK11195 which will be used as a marker of activated macrophages/microglia. The investigators will correlate [11C]PK11195 uptake with conventional measures of inflammation and neuronal integrity on high-resolution MRI.

SPMS subjects will have two baseline [11C]PK-11195 PET scans (separated by 24 to 72 hours, test-retest) and subsequent scans at 6, 12 and 24 months. SPMS Subjects will have brain MRI's at baseline, 6, 12 and 24 months.

Healthy Controls will have 2 baseline PET scans and one MRI.

DETAILED DESCRIPTION:
This is pilot study designed to determine the baseline and longitudinal regional-specific change in uptake of [11C]PK-11195 in subjects with secondary progressive multiple sclerosis (SPMS). Eighteen subjects with SPMS will be enrolled in the two-year study. Given low sample size, a stable treatment regimen is required to control for potential treatment effect. In addition, subjects must have been on current therapy for at least 6 months to ensure the measurement is reflective of true disease activity and not treatment effect. Thirteen age-matched healthy controls (HC) will be enrolled. The role of HC is to establish the variability or "noise" associated with the instrument (test-retest), which will ensure that PK uptake measured at any time point in MS is biologically relevant.

This proposal also includes a sub-study to validate a non-invasive quantification methodology for PK-PET. The most rigorous method, or gold standard, for quantifying PET data is based upon measuring the arterial input function. Measuring radioactivity within the arterial circulation requires arterial cannulation. Arterial cannulation is considered safe; however, is labor-intensive and often discourages subjects from participation. Image-derived input function (IDIF) is a method to calculate the input function without cannulation of the artery using the imaging data. Studies in human research volunteers are still required to compare the results obtained with classical arterial sampling and the IDIF. The current study will validate IDIF as a substitute for arterial sampling in this context. All healthy controls will undergo this validation process, which will include arterial and venous sampling. This validation is also required within subjects. Subjects will be given the option to participate in this validation stage.

Absolute Quantification of PK-PET (gold standard arterial sampling): Catheters will be placed in the radial artery for characterizing the plasma input function. This will make it possible to use a two tissue reversible plasma input (2T4k) model. Blood sampling will be acquired using both an online continuous blood sampling device as well as manually at discrete times (5, 10, 15, 20, 30, 40, 50 and 60 minutes post injection). The continuous sampling will be used to measure the activity concentrations of the whole blood, while the discrete manual sampling will be used to calculate the plasma concentration, and estimate the fraction of radioactive metabolites using HPLC. The total blood loss is estimated to be 8-10 tablespoons (120-150 mL, or about one third of the amount that volunteers donate to the Red Cross when giving blood). To generate the plasma input functions, the ratio of the plasma data to whole blood will be calculated for each manual blood sample and fitted through these points to a model with a one- or two-exponential function. Metabolite correction will be accomplished by multiplying the plasma curve with a function obtainable from a fit to the measured parent fraction. Venous blood will be similarly obtained for IDIF metabolic correction and utilized for validation against classic arterial sampling. The investigators will acquire up to 6 venous samples of 3 mL each with a 2 mL purge prior to each sample, for a total blood loss of 30 mL (one fluid ounce, or about 6.67% of the amount that volunteers donate to the Red Cross when giving blood).

Dynamic PET acquisition and processing: The data will be acquired in list mode to facilitate processing at any dynamic framing rate.

Innate immunity is recognized as a major cause of tissue injury in central nervous system (CNS) disease. In this study the investigators will specifically quantify the innate immune inflammatory burden in a cohort of secondary progressive multiple sclerosis (SPMS) subjects. Our hypothesis is that the innate immune response is heightened in SPMS as compared to healthy controls (HC's) and this activity increases over time and correlates with ongoing neuronal loss and disability. The investigators will test this hypothesis by using highly specific molecular imaging techniques, specifically PET, in conjunction with high field MRI. The investigators will utilize the PET radioligand [11C]1533; PK11195 which binds to the translocator protein 18 kDa (TSPO) on activated macrophages/microglia. The investigators will correlate [11C]PK11195 uptake with conventional measures of inflammation and neuronal integrity on high-resolution MRI.

MS is a chronic inflammatory disease of central nervous system characterized by focal T cell and macrophage infiltrates associated with demyelination. The primary innate immune cells in MS consist of infiltrating macrophages/monocytes and resident microglia. Cells of the innate immune system are effector cells that function to cause CNS injury both through direct effects on neighboring cells, such as oligodendrocytes, and through generation of soluble proinflammatory mediators that have distant effects on cells, such as neurons. The innate immune inflammatory is thus sufficient to explain focal injury and diffuse injury. In the majority of subjects, MS begins as a relapsing-remitting course but eventually evolves to a state of progressive decline in disability. Focal inflammatory demyelinating lesions are the predominant pathological findings in the subjects with relapsing disease whereas diffuse axonal injury with microglial activation has been found to be the hallmark of progressive disease.1 Microglial activation itself occurs either as a response to CNS injury for example as in Wallerian degeneration, or in response to signals from other inflammatory cells including macrophages and lymphocytes.

Activated microglia and infiltrating macrophages express TSPO (previously referred to as the peripheral benzodiazepine receptor) which can be detected with radioligand [11C]PK-111952.

Determination of the significance of any [11C]PK-11195 uptake within a cohort of MS subjects would require a correlation with HC¿s to ensure the observation is a valid measurement of disease activity.

The MS subjects will also have two baseline [11C]PK-11195 PET scans (separated by 24 to 72 hours, test-retest) to measure disease related intra-individual variability and will have subsequent scans at 6, 12 and 24 months. Baseline test-retest [11C]PK-11195 PET uptake between MS subjects and HC's will be compared to ensure minimal disease-related variability and to ensure our baseline and subsequent longitudinal measurements in MS subjects have met a level of biological significance. One baseline brain MRI is required for HC and MS subjects. Subjects will have brain MRI's at 6, 12 and 24 months.

Objective: Aim 1: To quantify level of activity and dynamic change in the innate immune inflammatory burden over the course of two years in a cohort of SPMS subjects.

Primary objective: Measure the level of baseline and change of whole brain uptake of [11C]PK-11195 at 6, 12 and 24 months in SPMS subjects.

Objectives:

* To correlate the change in T2-hyperintense lesion volume at 6,12 and 24 months of with whole brain uptake of [11C]PK-11195 on PET (at the 6,12 and 24 months) in SPMS subjects.
* To correlate the change of conventional MRI measures of neuronal integrity (Gray Matter Fraction, White Matter Fraction, whole brain volume, T1-hypointense lesion volume) at 6,12 and 24 months with whole brain PET uptake of [11C]PK-11195 (at the 6,12 and 24 months) in SPMS subjects.
* To correlate the change in whole brain PET uptake of [11C]PK-11195 (at the 6,12 and 24 months) and level in disability, as measured by a change in EDSS at 6, 12, and 24 months in SPMS subjects.

ELIGIBILITY:
Inclusion Criteria:

* Subjects age 18-80
* Secondary progressive MS subjects either untreated or on consistent treatment for six-months prior to enrollment
* Norman Controls

Exclusion Criteria:

* Subjects pregnant or woman of child-bearing age not utilizing effective birth control
* Primary progressive MS subjects
* Relapsing remitting MS subjects
* Unstable SPMS subject for which treatment change within the 24 months is likely

Age-Healthy controls will be excluded if have any of the following medical conditions:

* Any central nervous system disorder
* Any systemic auto-immune disorder
* Pregnant or woman of child-bearing age not utilizing effective birth control

Subjects will be withdrawn from the study if treatment is changed during the 24-month study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Approximately 36 subjects (with SPMS and controls) including screen failures will be enrolled regardless of gender
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2014-07; Primary Completion 2020-12 (Actual); Study Completion 2020-12 (Actual)

PRIMARY OUTCOMES:
Measure the level of baseline and change of whole brain uptake of [11C]PK-11195 at 6, 12 and 24 months in SPMS subjects. | 24 months

SECONDARY OUTCOMES:
To correlate the change in T2-hyperintense lesion volume at 6,12 and 24 months of with whole brain uptake of [11C]PK-11195 on PET (at the 6,12 and 24 months) in SPMS subjects. | 24 months
To correlate the change of conventional MRI measures of neuronal integrity (Gray Matter Fraction, White Matter Fraction, whole brain volume, T1-hypointense lesion volume) at 6,12 and 24 months with whole brain PET uptake of [11C]PK-11195 (at the 6,12 and | 24 months
To correlate the change in whole brain PET uptake of [11C]PK-11195 (at the 6,12 and 24 months) and level in disability, as measured by a change in EDSS at 6, 12, and 24 months in SPMS subjects. | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Susan Gauthier, DO, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medical College, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No